CLINICAL TRIAL: NCT00805467
Title: An Open-Label, Multicenter Extension Study to Evaluate the Safety of R935788 in Patients With Rheumatoid Arthritis Who Have Completed the Treatment Phase of a Rigel-Sponsored R935788 Study
Brief Title: Open-Label, Multicenter Extension Study for Patients Completing Treatment Phase of a Rigel-Sponsored R935788 Studies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-935788-012; D4300C00021
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): R935788 50 mg tablet, orally, twice-a-day
  Interventions: Drug: Fostamatinib Disodium (R935788)
- 2 (Experimental): R935788 100 mg tablet, orally, twice-a-day
  Interventions: Drug: Fostamatinib Disodium (R935788)
- 3 (Experimental): R935788 100 mg tablet, orally, once-a-day
  Interventions: Drug: Fostamatinib Disodium (R935788)
- 4 (Experimental): R935788 150 mg tablet, orally, once-a-day
  Interventions: Drug: Fostamatinib Disodium (R935788)

INTERVENTIONS:
Drug: Fostamatinib Disodium (R935788) — 50 mg PO BID; 100 mg PO BID; 100 mg PO QD; 150 mg tablet PO QD
  Other Names: R935788

SUMMARY:
The purpose of this new research study is to gain additional information about how safe and effective R935788 is over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent by signing an IRB/EC-approved Informed Consent Form (ICF) prior to admission to this study
* Patients who are being treated in Study C-788-006X
* Patients who completed Studies C-788-010 or C-788-011 and did not withdraw due to adverse events
* Patients who withdrew from Study C-788-010 at Month 4 or Month 5 because of a pre-defined lack of efficacy
* Females of childbearing potential must be fully informed of the potential for R788 to adversely affect the fetus and, if sexually active, must agree to use a well established method of birth control during the study (oral contraceptive, mechanical barrier, long acting hormonal agent). These patients must not be lactating and must have a negative pregnancy test at the time of entry and at each laboratory determination.

Exclusion Criteria:

* The patient has a history of, or a concurrent, clinically significant illness, medical condition (other than arthritis) or laboratory abnormality that, in the Investigator's opinion, could affect the conduct of the study. Specifically, excluded are patients with the following:

  1. unresolved Grade 2 or greater toxicity in a RA protocol studying R788
  2. uncontrolled or poorly controlled hypertension;
  3. recent (within past 2 months) serious surgery or infectious disease;
  4. recent history (since enrollment in prior R788 study) of, or treatment for, a malignancy other than non-melanomatous skin cancer, or any history of lymphoma;
  5. known to be positive for Hepatitis B, Hepatitis C, HIV or Tuberculosis;
  6. interstitial pneumonitis or active pulmonary infection;
  7. known laboratory abnormalities: ALT > 1.2 x ULN, creatinine >1.5x ULN, an ANC <2,500/mm3 or 2.5 x 109/L, lymphocyte count < 600/mm3 or 0.6 x 109L, Hgb < 9 g/dL or 5 mmol/L, platelet count <125,000/mm3 or 125 x 109/L are excluded.
* The patient has a history of substance abuse, drug addiction or alcoholism. Patients may consume up to 4 units of alcohol per week; however, alcohol should be avoided in the 72 hours prior to lab assessments. Patients who cannot reliably comply with this should be excluded. A unit of alcohol is defined as the following: Beer = 12 oz or 355 mL; wine = 5 oz or 148 mL; sweet dessert wine = 3 oz or 89 mL; 80 proof distilled spirits = 1.5 oz or 44 mL.
* The patient is unable to report for clinical and laboratory monitoring as per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2008-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, PhD, Study Director — AstraZeneca
Locations (76):
- United States (35):
  - Research Site, La Jolla, California
  - Research Site, Palm Desert, California
  - Research Site, Palo Alto, California
  - Research Site, San Diego, California
  - Research Site, Santa Maria, California
  - Research Site, Hamden, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Aventura, Florida
  - Research Site, Boca Raton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, South Miami, Florida
  - Research Site, Venice, Florida
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, South Bend, Indiana
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Cumberland, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Lansing, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Roslyn, New York
  - Research Site, Smithtown, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Mayfiled Village, Ohio
  - Research Site, Erie, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Oklahoma City, Washington
  - Research Site, Spokane, Washington
- Belgium (3):
  - Research Site, Antwerp
  - Research Site, Ghent
  - Research Site, Liège
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Medellín
- Research Site, Bordeaux, France
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Würzburg
- Italy (2):
  - Research Site, Siena
  - Research Site, Udine
- Mexico (9):
  - Research Site, Chihuahua City
  - Research Site, Cuernava
  - Research Site, Del. Cuauhtemoc
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, Mexcio
  - Research Site, México
  - Research Site, Morelia
  - Research Site, San Luis Potosí City
- Peru (2):
  - Research Site, Jesus Maria
  - Research Site, Lima
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bytom
  - Research Site, Elblag
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Torun
  - Research Site, Wroclaw
  - Research Site, Zyrardów
- Romania (5):
  - Research Site, Brailari
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Sf. Gheorghe
  - Research Site, Sibiu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 624 patients were enrolled: 1, 59, 183 & 381 were allocated to the 50mg twice daily (bid), 100 mg once daily (qd), 150 mg qd and 100 mg bid groups, respectively. As this was a long-term extension study no specific end date was given. Patients who were ongoing when the study was terminated are shown as completers.
Pre-assignment Details: Treatments were assigned according to those given in the qualifying studies. All patients received investigational product.
Groups:
- Fostamatinib 50 mg Bid; Fostamatinib 100 mg qd; Fostamatinib 150 mg qd; Fostamatinib 100 mg Bid: Oral treatment
Period: Overall Study
Arm/Group | Fostamatinib 50 mg Bid | Fostamatinib 100 mg qd | Fostamatinib 150 mg qd | Fostamatinib 100 mg Bid
Started | 1 (Patients who received treatment) | 59 (Patients who received treatment) | 183 (Patients who received treatment) | 381 (Patients who received treatment)
Enrolled But Did Not Receive Treatment | 0 | 0 | 0 | 0
Completed | 1 (Ongoing when study terminated) | 25 (Ongoing when study terminated) | 80 (Ongoing when study terminated) | 144 (Ongoing when study terminated)
Not Completed | 0 | 34 | 103 | 237
Not completed — Lack of Efficacy | 0 | 8 | 13 | 86
Not completed — Lost to Follow-up | 0 | 1 | 7 | 21
Not completed — Withdrawal by Subject | 0 | 6 | 45 | 50
Not completed — Protocol Violation | 0 | 3 | 0 | 5
Not completed — Adverse Event | 0 | 13 | 26 | 57
Not completed — Death | 0 | 2 | 7 | 5
Not completed — Physician Decision | 0 | 1 | 2 | 6
Not completed — Not reported | 0 | 0 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib 50 mg Bid | Fostamatinib 100 mg qd | Fostamatinib 150 mg qd | Fostamatinib 100 mg Bid | Total
Number analyzed (Participants) | 1 | 59 | 183 | 381 | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (NA) — Standard deviation cannot be defined for a single patient. | 51.4 (11.15) | 51.7 (13.32) | 53.8 (12.36) | 53.0 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 53 | 157 | 324 | 535
  Male | 0 | 6 | 26 | 57 | 89
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 0 | 18 | 88 | 184 | 290
  Black | 1 | 1 | 6 | 14 | 22
  Hispanic | 0 | 40 | 88 | 179 | 307
  Asian | 0 | 0 | 0 | 2 | 2
  Other | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had at Least 1 Treatment Emergent Adverse Event in Any Category
Description: AE = adverse event, bid = twice daily, IP = investigational product, qd = once daily, SAE = serious adverse event
Time Frame: Entry in extension to end of study, up to a maximum of 5 years. (Variable by subject - median duration of 3 years)
Population: The full analysis set includes those patients who received at least 1 dose of investigational product, and were summarised according to treatment first received in this study (intention-to-treat principle).
Measure: Number; unit: % of patients
Arm/Group | Fostamatinib 50 mg Bid | Fostamatinib 100 mg qd | Fostamatinib 150 mg qd | Fostamatinib 100 mg Bid
Number analyzed (Participants) | 1 | 59 | 183 | 381
% of patients
  Any AE | 100 | 91.5 | 90.7 | 88.7
  Any fatal AE | 0 | 1.7 | 3.8 | 1.6
  Any SAE (including fatal AEs) | 100 | 3.4 | 18.6 | 20.2
  Any AE leading to termination of study therapy | 0 | 22.0 | 16.4 | 15.2

2. Secondary Outcome: DAS28-CRP Score
Description: The Disease Activity Score 28 using C-Reactive Protein (DAS28-CRP) is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). These measures are then fed into a complex mathematical formula to produce the overall DAS on a scale from 1 to 10, where scores greater than 5.1 are considered to indicate active disease, scores less than 3.2 are considered to indicate with well controlled disease, and scores less than 2.6 are considered to indicate remission. bid = twice daily, CRP = C-reactive protein, DAS28 = Disease Activity Score based on a 28 joint count, n/a = not applicable, qd = once daily
Time Frame: 3 years
Population: Number of participants are those with baseline data. Baseline defined at entry into qualifying study or at entry into this study if more than 14 days since last dose in qualifying study. As no imputation was applied, the numbers at subsequent visits are lower.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fostamatinib 50 mg Bid | Fostamatinib 100 mg qd | Fostamatinib 150 mg qd | Fostamatinib 100 mg Bid
Number analyzed (Participants) | 1 | 55 | 181 | 374
scores on a scale
  Baseline (n=1, 55, 181, 374) | 5.27 (NA) — Standard deviation cannot be defined for a single patient. | 5.34 (1.123) | 5.31 (1.162) | 5.36 (1.259)
  Quarter 4 (n=1, 41, 136, 254) | 2.00 (NA) — Standard deviation cannot be defined for a single patient. | 3.57 (1.408) | 3.46 (1.282) | 3.44 (1.453)
  Quarter 8 (n=1, 33, 114, 201) | 2.92 (NA) — Standard deviation cannot be defined for a single patient. | 3.43 (1.412) | 3.25 (1.290) | 3.35 (1.484)
  Quarter 12 (n=1, 30, 94, 174) | 2.31 (NA) — Standard deviation cannot be defined for a single patient. | 3.36 (1.376) | 3.07 (1.055) | 3.27 (1.373)

3. Secondary Outcome: HAQ-DI Score
Description: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is calculated by summing the category scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygeine, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability. A HAQ-DI response is a reduction from baseline in HAQ-DI greater than or equal to the minimally important difference (0.22). BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Fostamatinib 50 mg Bid | Fostamatinib 100 mg qd | Fostamatinib 150 mg qd | Fostamatinib 100 mg Bid
Number analyzed (Participants) | 1 | 56 | 181 | 376
Scores on a Scale
  Baseline (n=1, 56, 181, 376) | 1.25 (NA) — Standard deviation cannot be defined for a single patient | 1.50 (0.735) | 1.46 (0.707) | 1.46 (0.715)
  Quarter 4 (n=1, 41, 138, 254) | 0.57 (NA) — Standard deviation cannot be defined for a single patient | 1.00 (0.677) | 1.07 (0.726) | 0.99 (0.722)
  Quarter 8 (n=1, 33, 107, 201) | 0.43 (NA) — Standard deviation cannot be defined for a single patient | 1.00 (0.657) | 1.02 (0.720) | 0.95 (0.703)
  Quarter 12 (n=1, 30, 94, 176) | 0.38 (NA) — Standard deviation cannot be defined for a single patient | 1.01 (0.651) | 0.98 (0.718) | 0.96 (0.687)

ADVERSE EVENTS:
Arm/Group | 100 MG BID | 100 MG QD | 150 MG QD | 50 MG BID
Serious Adverse Events (participants affected / at risk) | 77/381 | 2/59 | 34/183 | 1/1
Other Adverse Events (participants affected / at risk) | 306/381 | 49/59 | 141/183 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 MG BID (N=381) | 100 MG QD (N=59) | 150 MG QD (N=183) | 50 MG BID (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANOPHTHALMITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRIC PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PANCREATITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS SOFT TISSUE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS HEPATITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSENTERY (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPIGLOTTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA MIGRANS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
GIARDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTED BITES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 6 (7) | 0 (0) | 3 (3) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BASOSQUAMOUS CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS INCOMPLETE (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
IMPLANTABLE DEFIBRILLATOR INSERTION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 MG BID (N=381) | 100 MG QD (N=59) | 150 MG QD (N=183) | 50 MG BID (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 24 (28) | 1 (1) | 13 (17) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 30 (34) | 5 (5) | 10 (13) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 11 (11) | 3 (3) | 5 (5) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (10) | 3 (3) | 3 (4) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 96 (151) | 20 (36) | 60 (93) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 8 (8) | 3 (4) | 3 (4) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 14 (15) | 5 (5) | 8 (8) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 27 (31) | 3 (4) | 11 (12) | 0 (0)
VOMITING (Gastrointestinal disorders) | 23 (27) | 5 (9) | 10 (11) | 0 (0)
CHEST PAIN (General disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 24 (34) | 3 (3) | 7 (8) | 0 (0)
BRONCHITIS (Infections and infestations) | 26 (38) | 3 (4) | 14 (20) | 0 (0)
INFLUENZA (Infections and infestations) | 36 (54) | 8 (15) | 18 (20) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 27 (31) | 3 (3) | 10 (12) | 0 (0)
PHARYNGITIS (Infections and infestations) | 16 (19) | 5 (6) | 5 (6) | 0 (0)
SINUSITIS (Infections and infestations) | 26 (37) | 3 (3) | 4 (4) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 51 (76) | 7 (8) | 20 (29) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 72 (125) | 12 (32) | 28 (45) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 27 (35) | 1 (1) | 11 (11) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 6 (10) | 0 (0) | 2 (5) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 35 (45) | 7 (8) | 15 (16) | 0 (0)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 (16) | 3 (3) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 (25) | 1 (2) | 10 (16) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 30 (35) | 3 (3) | 9 (11) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 16 (20) | 4 (5) | 5 (5) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 (10) | 3 (3) | 2 (2) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 38 (69) | 3 (6) | 10 (16) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 33 (49) | 4 (7) | 23 (35) | 0 (0)
HYPERTONIC BLADDER (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 2 (2) | 8 (9) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 9 (10) | 3 (3) | 8 (9) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 62 (82) | 10 (13) | 26 (31) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other